CLINICAL TRIAL: NCT07320573
Title: Evaluation of Pelvic Floor Muscle Strength in Women With Stress Urinary Incontinence Using Two Different EMG Methods
Brief Title: Evaluation of Pelvic Floor Muscle Strength in Women With Stress Urinary Incontinence
Status: Not yet recruiting | Type: Observational
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Esra BAYRAMOĞLU DEMİRDÖĞEN, LecTURER DOCTOR, Ahi Evran University Education and Research Hospital
Other Study IDs: KAEU-EBAYRAMOGLUD-004
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Floor Muscle Strength Measurement
MeSH Terms: interventions — Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- stress urinary incontinence: Pelvic floor muscle strength will be measured superficially, intravaginally, and digitally.
  Interventions: Device: Electromyography

INTERVENTIONS:
Device: Electromyography — Muscle strength values will be obtained using surface electrodes.

SUMMARY:
Pelvic floor muscle strength will be measured in women with stress urinary incontinence using superficial EMG, intravaginal EMG, and digital palpation. A 10-minute rest period will be given between each measurement, and the results will be recorded. Once all measurements are completed, any differences between the three measurements will be examined.

DETAILED DESCRIPTION:
Pelvic floor muscle strength will be assessed by vaginal palpation in the women included in the study. Then, patients will be placed in a hook position for EMG measurement. For superficial measurement, electrodes will be placed on the levator ani muscle on either side, and then the first assessment will be performed in 3 trials consisting of 5 seconds of contraction followed by 5 seconds of rest, and the second assessment in 3 trials consisting of 2 seconds of contraction followed by 5 seconds of rest.

Measurement with an intervaginal electrode will also be performed in the supine hook position, using a passive electrode and an active vaginal probe. Lubricant gel will be applied to the vaginal probe before insertion into the vagina, and the passive electrode will be placed on the inner surface of the right thigh (adductor muscle group). Two different protocols will be used for assessment. The first assessment will consist of 3 trials of 5 seconds of contraction followed by 5 seconds of rest, and the second assessment will consist of 3 trials of 2 seconds of contraction followed by 5 seconds of rest. A 10-minute rest period will be included between measurements. The ICIQ-SF questionnaire will also be used to determine the type and degree of incontinence. Participants will be asked to answer the questions considering the last two weeks. A score will then be assigned.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having stress urinary incontinence
* Being willing to participate in the study

Exclusion Criteria:

* Unwillingness to continue working
* Presence of a neurological disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with stress urinary incontinence
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-14 (Estimated)

PRIMARY OUTCOMES:
pelvic floor muscle strength | day 1
  muscle strength and endurance durations

CONTACTS AND LOCATIONS:
Locations (1):
- Kirşehir Ahi Evran University Physical Therapy and Rehabilitation Hospital, Kırşehir, Centre, Turkey (Türkiye)